CLINICAL TRIAL: NCT03909100
Title: International CoolSculpting: Prospective, Multi-Country, Study to Evaluate Patient Satisfaction for Non-Invasive Fat Reduction in Abdomen and/or Flanks (iCOOL)
Brief Title: International CoolSculpting: Study to Evaluate Patient Satisfaction for Non-Invasive Fat Reduction in Abdomen and/or Flanks (iCOOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO-MA-PLS-0602
Record Dates: First submitted 2019-03-18; First posted 2019-04-09 (Actual); Results first posted 2021-03-22 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Non-invasive Fat Reduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CoolSculpting® System (Experimental): Participants received up to two CoolSculpting® treatment sessions for the abdomen, flanks or both 8 weeks apart. A treatment session was comprised of timed segments of cooling (treatment cycles) followed by 2 minutes of manual massage. Up to 12 cycles per treatment session were performed at the investigator's discretion.
  Interventions: Device: CoolSculpting® System

INTERVENTIONS:
Device: CoolSculpting® System — A treatment session is comprised of timed segments of cooling (treatment cycles) followed by 2 minutes of manual massage.

SUMMARY:
This study aims to generate data that conveys participant's experiences such as their overall satisfaction with the CoolSculpting® treatment for their belly and love handles. By doing this, the study will provide insights for doctors to better inform participants about the expected outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participant has clearly visible fat in the flanks and/or abdomen, which in the investigator's opinion, may benefit from the treatment.
* Participant has not had weight change fluctuations exceeding 4.5 kg (or 5% of body weight) in the preceding month.
* Participant has a body mass index (BMI) of 18.5 to 30. A BMI is defined as weight in kilograms divided by height in meters squared (kg/m2).
* Participant agrees to maintain weight (ie, within 5% of body weight) by not making any changes in diet or exercise routine during the course of the study.
* Participant agrees to have photographs taken of the treatment area(s) during the scheduled time periods.

Exclusion Criteria:

* Participant has had liposuction, or another surgical procedure(s) or mesotherapy in area of intended treatment.
* Participant has had a non-invasive fat reduction and/or body contouring procedure in the area(s) of intended treatment within the past 12 months.
* Participant needs to administer, or has a known history of subcutaneous injections into the area(s) of intended treatment (eg, cortisone, heparin, insulin) within the past 6 months.
* Participant is pregnant or intending to become pregnant.
* Participant is lactating or has been lactating in the past 6-9 months.
* Participant is unable or unwilling to comply with study requirements.
* Participant is currently enrolled in a clinical study of any unapproved investigational device, investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Participant has an active implanted device such as a pacemaker, defibrillator, or drug delivery system or any other metal containing implant.
* Participant with known history of cryoglobulinemia, cold agglutinin disease, or paroxysmal cold hemoglobinuria.
* Participant with known sensitivity to cold or has any condition with a known response to cold exposure that limits blood flow to the skin such as cold urticaria or Raynaud's disease, or Chilblains (pernio).
* Participant with known sensitivity or allergy to fructose, glycerin, isopropyl alcohol, or propylene glycol.
* Participant with impaired peripheral circulation in the area to be treated
* Participant with neuropathic disorders such as post-herpetic neuralgia or diabetic neuropathy.
* Participant with impaired skin sensation.
* Participant with open or infected wounds.
* Participant with bleeding disorders, or concomitant use of blood thinners, or is taking any medication that in the investigator's opinion may increase the participant's risk of bruising.
* Participant with recent surgery or scar tissue in the area to be treated.
* Participant has history of hernia in or adjacent to the treatment area(s) site.
* Participant with skin conditions such as eczema, dermatitis, or rashes in the area to be treated.
* Participant has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Participant is taking or has taken diet pills or supplements within the past 6 months.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the participant's response or the integrity of the data or would pose an unacceptable risk to the participant.
* Participant diagnosed with fibrosis.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Jo, Study Director — Allergan
Locations (7):
- Australia (2):
  - Sandhurt Plastic Surgery, Bendigo, Victoria
  - Academy Face and Body, Subiaco, Western Australia
- Vancouver Laser & Skin Care Centre, Vancouver, British Columbia, Canada
- Singapore (2):
  - Halley Medical Aesthetics, Singapore
  - Dr Benjamin Yim Clinical Aesthetics and Laser Centre, Singapore
- United Kingdom (2):
  - Revere Riverside Ltd, Northwood, Middlesex
  - Revere Clinics, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CoolSculpting® System
Started | 120
Safety Population (All participants who had at least 1 of the treatment procedures conducted.) | 112
Received Treatment in Session 2 | 107
Evaluable Population (Evaluable Population included all participants who signed the informed consent form (ICF), had at least 1 of the procedures conducted, and also reported the Cryolipolysis Satisfaction Questionnaire (CSQ) Item 1 at 12 weeks after the final treatment (measured at Week 12 for participants who received 1 treatment session and at Week 20 for participants who received 2 treatment sessions).) | 106
Completed | 105
Not Completed | 15
Not completed — Protocol Deviation | 2
Not completed — Technical Problems | 4
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Not completed — Reason not Specified | 4

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who had at least 1 of the treatment procedures conducted.
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48
  Black | 1
  Asian - Chinese | 51
  Asian - Korean | 1
  Asian, Other | 9
  Arab/Middle Eastern | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Reported "Satisfied" or "Very Satisfied" on Cryolipolysis Satisfaction Questionnaire (CSQ) Item #1 Overall
Description: The CSQ is a 4-item Patient-reported Outcome (PRO) instrument that measures the participant's satisfaction with CoolSculpting® treatment of the flank, abdomen or both. Participants rated their satisfaction by answering CSQ Item 1="Rate your overall satisfaction with the fat reduction procedure on the treated area" using the following scale: Very satisfied, Satisfied, Neither satisfied nor dissatisfied, Dissatisfied or Very dissatisfied.
Time Frame: 12 weeks after the final treatment session (measured at Week 12 for participants who received 1 treatment session or Week 20 for 2 treatment sessions)
Population: Evaluable Population included all participants who signed the ICF, had at least 1 of the procedures conducted, and also reported the CSQ Item 1 at 12 weeks after the final treatment (measured at Week 12 for participants who received 1 treatment session and at Week 20 for participants who received 2 treatment sessions).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 106
percentage of participants | 89.6 [83.8 to 95.4]

2. Secondary Outcome: Percentage of Participants Who Reported "Satisfied" or "Very Satisfied" on CSQ Item #1 in Treated Area(s)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Evaluable Population included all participants who signed the ICF, had at least 1 of the procedures conducted, and also reported the CSQ Item 1 at 12 weeks after the final treatment (measured at Week 12 for participants who received 1 treatment session and at Week 20 for participants who received 2 treatment sessions). Number analyzed are the number of participants with evaluable data for given category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 106
percentage of participants
  Abdomen | 87.1 [80.6 to 93.7]
  Flanks | 93.1 [88.1 to 98.0]
  Abdomen and Flanks: number analyzed (Participants) | 96
  Abdomen and Flanks | 89.6 [83.5 to 95.7]

3. Secondary Outcome: Percentage of Participants Who Received 1 or 2 Treatments Who Reported "Satisfied" or "Very Satisfied" on CSQ Item #1 by Number of Treatment Cycles
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 106
percentage of participants
  24 Treatment Cycles: number analyzed (Participants) | 51
  24 Treatment Cycles | 92.2 [84.8 to 99.5]
  22 Treatment Cycles: number analyzed (Participants) | 1
  22 Treatment Cycles | 100.0 [100.0 to 100.0]
  21 Treatment Cycles: number analyzed (Participants) | 1
  21 Treatment Cycles | 100.0 [100.0 to 100.0]
  20 Treatment Cycles: number analyzed (Participants) | 4
  20 Treatment Cycles | 100.0 [100.0 to 100.0]
  18 Treatment Cycles: number analyzed (Participants) | 5
  18 Treatment Cycles | 80.0 [44.9 to 100.0]
  17 Treatment Cycles: number analyzed (Participants) | 1
  17 Treatment Cycles | 100.0 [100.0 to 100.0]
  16 Treatment Cycles: number analyzed (Participants) | 13
  16 Treatment Cycles | 92.3 [77.8 to 100.0]
  15 Treatment Cycles: number analyzed (Participants) | 3
  15 Treatment Cycles | 100.0 [100.0 to 100.0]
  14 Treatment Cycles: number analyzed (Participants) | 6
  14 Treatment Cycles | 66.7 [28.9 to 100.0]
  13 Treatment Cycles: number analyzed (Participants) | 1
  13 Treatment Cycles | 100.0 [100.0 to 100.0]
  12 Treatment Cycles: number analyzed (Participants) | 10
  12 Treatment Cycles | 80.0 [55.2 to 100.0]
  11 Treatment Cycles: number analyzed (Participants) | 1
  11 Treatment Cycles | 100.0 [100.0 to 100.0]
  10 Treatment Cycles: number analyzed (Participants) | 2
  10 Treatment Cycles | 100.0 [100.0 to 100.0]
  9 Treatment Cycles: number analyzed (Participants) | 2
  9 Treatment Cycles | 100.0 [100.0 to 100.0]
  7 Treatment Cycles: number analyzed (Participants) | 1
  7 Treatment Cycles | 0 [0 to 0]
  6 Treatment Cycles: number analyzed (Participants) | 2
  6 Treatment Cycles | 100.0 [100.0 to 100.0]
  5 Treatment Cycles: number analyzed (Participants) | 1
  5 Treatment Cycles | 100.0 [100.0 to 100.0]
  2 Treatment Cycles: number analyzed (Participants) | 1
  2 Treatment Cycles | 100.0 [100.0 to 100.0]

4. Secondary Outcome: Percentage of Participants by Body Mass Index (BMI) Categories Who Reported "Satisfied" or "Very Satisfied" on CSQ Item #1
Description: The CSQ is a 4-item Patient-reported Outcome (PRO) instrument that measures the participant's satisfaction with CoolSculpting® treatment of the flank, abdomen or both. Participants rated their satisfaction by answering CSQ Item 1="Rate your overall satisfaction with the fat reduction procedure on the treated area" using the following scale: Very satisfied, Satisfied, Neither satisfied nor dissatisfied, Dissatisfied or Very dissatisfied. Participants were analyzed based on BMI ranges from 18.5 to < 25.0 and 25.0 to < 30.0. BMI was defined as weight in kilograms divided by height in meters squared (kg/m^2).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 106
percentage of participants
  BMI 18.5 - < 25: number analyzed (Participants) | 52
  BMI 18.5 - < 25 | 88.5 [79.8 to 97.1]
  BMI 25 - ≤ 30: number analyzed (Participants) | 54
  BMI 25 - ≤ 30 | 90.7 [83.0 to 98.5]

5. Secondary Outcome: Change From Baseline in Volume of Fat as Measured by 3 Dimensional (3D) Photography
Description: Change in the volume of fat was assessed by a 3D stereoscopic camera which was used to generate a 3D image of the body, allowing quantification of the abdomen and flank areas. A 2-step 3D matching algorithm process was used, to identify the change of volume in milliliters (mL).
Time Frame: Baseline to 8 Weeks post-Treatment 1 and 12 Weeks post-Final Treatment 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 106
mL
  Change from Baseline at 8 Weeks Post-Treatment Session 1: number analyzed (Participants) | 96
  Change from Baseline at 8 Weeks Post-Treatment Session 1 | -149.1 (280.61)
  Change from Baseline at 12 Weeks Post-Final Treatment: number analyzed (Participants) | 97
  Change from Baseline at 12 Weeks Post-Final Treatment | -264.8 (411.36)

6. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, users, or other persons, if related to the investigational medical device. A SAE is any AE, that is fatal, life threatening, requires hospitalization or results in prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. A TEAE is defined as any new adverse event or worsening of an existing condition after initiation of treatment.
Time Frame: First treatment to Follow-up/Exit Visit (Week 12 +/- 14 days for those participants who received 1 treatment and Week 20 +/- 14 days for those participants who received 2 treatments)
Population: Safety Population included all participants who had at least 1 of the treatment procedures conducted.
Measure: Number; unit: percentage of participants
Groups:
- CoolSculpting®: Treatment Session 1: Participants who received one CoolSculpting® treatment session for the abdomen, flanks or both. A treatment session was comprised of timed segments of cooling (treatment cycles) followed by 2 minutes of manual massage. Up to 12 cycles per treatment session were performed at the investigator's discretion.
- CoolSculpting®: Treatment Session 2: Participants who received a second CoolSculpting® treatment session for the abdomen, flanks or both 8 weeks after the first session. A treatment session was comprised of timed segments of cooling (treatment cycles) followed by 2 minutes of manual massage. Up to 12 cycles per treatment session were performed at the investigator's discretion.
Arm/Group | CoolSculpting®: Treatment Session 1 | CoolSculpting®: Treatment Session 2
Number analyzed (Participants) | 112 | 107
percentage of participants
  TEAE | 14.3 | 10.3
  SAE | 0.0 | 0.9

7. Secondary Outcome: Percentage of Participants With Adverse Device Effects (ADEs) and Serious Adverse Device Effects (SADEs)
Description: An ADE was defined in accordance with ISO 14155 as an AE related to the use of an investigational medical device or defined as AE with a reasonable possibility (Possible, Probable, or Causal relationship) that the device caused the event. SADE is an ADE that might have led to any SAE consequences if a suitable action had not been taken or intervention had not been made.
Time Frame: as for outcome 6
Population: Safety Population included all participants who had at least 1 of the treatment procedures conducted.
Measure: Number; unit: percentage of participants
Arm/Group | CoolSculpting®: Treatment Session 1 | CoolSculpting®: Treatment Session 2
Number analyzed (Participants) | 112 | 107
percentage of participants
  ADE | 14.3 | 9.3
  SADE | 0 | 0

ADVERSE EVENTS:
Time Frame: First treatment to Follow-up/Exit Visit (Week 12 +/- 14 days for those participants who received 1 treatment and Week 20 +/- 14 days for those participants who received 2 treatments)
Description: Safety Population included all participants who had at least 1 of the treatment procedures conducted. AEs are reported separately for each of the two treatment sessions.
Arm/Group | CoolSculpting®: Treatment Session 1 | CoolSculpting®: Treatment Session 2
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/112 | 1/107
Other Adverse Events (participants affected / at risk) | 10/112 | 1/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | CoolSculpting®: Treatment Session 1 (N=112) | CoolSculpting®: Treatment Session 2 (N=107)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/83 | 1/79 — Number of participants at risk are female participants as this adverse event is specific to females.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CoolSculpting®: Treatment Session 1 (N=112) | CoolSculpting®: Treatment Session 2 (N=107)
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT03909100/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03909100/SAP_001.pdf